CLINICAL TRIAL: NCT02630342
Title: The Use of a Mock MRI Scanner for Reducing the Use of Anesthesia in Children Undergoing Clinical MRI Scans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Alberta Children's Hospital (Other)
Responsible Party: Principal Investigator, David Lardner, Co-Prinicpal Investigator, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REB-15-368
Record Dates: First submitted 2015-12-09; First posted 2015-12-15 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Magnetic Resonance Imaging
Keywords: Mock Scanner; Child Life Specialist; Patient Preparation; Child, Preschool; Child; Anxiety; Human; Anesthesia, General
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1: preparation materials only (Experimental): This group will receive preparation materials for a clinical MRI scan. These include links to online videos about MRI, audio files with scanner noises, and a childrens book about MRI scan. Preparation for this group will occur only at home.
  Interventions: Behavioral: Preparation materials
- Group 2: Materials with review (Experimental): This group will receive in preparation for a clinical MRI scan links to online videos about MRI, audio files with scanner noises, and a childrens book about MRI scan. Preparation for this group will occur at home and include a visit with research team to review preparation materials with the research team
  Interventions: Behavioral: Preparation materials; Behavioral: Review Preparation Materials
- Group 3: Mock MRI scanner (Experimental): This group will receive the same materials as training group 1. In addition they will attend the mock scanner where the research team will utilise a mock MRI scanner to practice lying down in a scanner, staying still , wearing headphones and watching a movie/video on the mirror system.
  Interventions: Behavioral: Mock MRI scanner; Behavioral: Preparation materials
- Neuro-oncology retrospective controls (No Intervention): A retrospective control group of neuro-oncology patients from the 3 years prior to the study initiation. This group will be used to determine the age at which patients were able to complete a diagnostic MRI without GA
- Neuro-oncology prospective (Experimental): Child life specialist preparation will be provided to these patients. This preparation for Diagnostic MRI scanning in which utilise the Mock MRI scanner as preparation for the scan.
  Interventions: Behavioral: Mock MRI scanner; Behavioral: Child Life Specialist preparation

INTERVENTIONS:
Behavioral: Mock MRI scanner — Using a mock scanner for preparation for MRI
  Arms: Group 3: Mock MRI scanner; Neuro-oncology prospective
Behavioral: Preparation materials — links to online videos about MRI, audio files with scanner noises, and a childrens book about MRI scan.
  Arms: Group 1: preparation materials only; Group 2: Materials with review; Group 3: Mock MRI scanner
Behavioral: Child Life Specialist preparation — Child Life Therapist will coordinate the prepartion of the child
  Arms: Neuro-oncology prospective
Behavioral: Review Preparation Materials — Review of preparation materials at the hospital with member of research team
  Arms: Group 2: Materials with review

SUMMARY:
Diagnostic Magnetic Resonance (MR) imaging procedures can be stressful for children and parents. Patients must lie still during the procedure to provide diagnostic quality images. Children <7 years are often sedated or given general anesthesia (GA) for imaging procedures. The high cost of GA and its associated risks motivate the search for alternatives. The overall goal of this study is to systematically investigate whether training on the mock MR scanner reduces the need for GA during Magnetic Resonance Imaging (MRI) scans in children.

160 participants scheduled for diagnostic MRI scans at Alberta Children's Hospital (ACH) will be recruited to undergo different training methods for MRI scanning. Group 1 will be sent links to online videos about MRI, audio files with scanner noises, and a children's book about MR scans, to prepare at home. Group 2 will receive training materials and visit the ACH to review them with the research team, but will not use the mock scanner. Group 3 will receive training materials and visit the ACH for training on the mock MR scanner. Visits to the mock scanner for Group 3 will include practice lying down, staying still, wearing headphones, and watching a movie on the mirror system. During and after training sessions, the investigators will collect data on total time spent preparing (mock scanner or other), the child's feelings of stress/worry before and after visit, and head motion during mock MRI session (if applicable).

Subjects will be scheduled for a clinical scan without GA and a follow-up clinical scan with GA (to be cancelled if the first scan is successful). Scan success will be determined by a radiologist. Measures of scan success, quality ratings for each scan, children's feelings of stress/worry related to the MRI, and saliva samples to measure cortisol and salivary alpha amylase, will be gathered at the clinical scan. An ANOVA will be used to compare different training groups.

A clinical group of 35 neuro-oncology patients aged 3-7 years of age that undergo frequent MRI scans will also undergo staged preparation by child life specialists using the mock scanner. The age at which they are able to complete MRI without general anesthesia will be compared with a retrospective control group in the 3 years prior. Measures to be used for this group are the same (with the exception of saliva samples). T test and Kaplan- Meier analysis will be used to compare age at which MRI can be performed awake.

DETAILED DESCRIPTION:
Diagnostic MR procedures can be scary and stressful for children and parents. Because patients must lie still during the procedure to provide diagnostic quality images, young children (typically <7 years) and others not expected to comply are often sedated or given general anesthesia (GA) for imaging procedures. However, the high cost of GA and its associated risks motivate the search for alternatives. Previous reports demonstrate that preparation (including using a mock MR scanner) reduces anxiety and increases compliance for clinical and research MRI procedures without GA. However, systematic studies of the advantages of a mock MR scanner versus other training methods are lacking. Furthermore, while reducing the use of GA is desirable, repeated unsuccessful scanning procedures are also costly, so identifying factors that predict success for diagnostic MR procedures is important to effectively allocate resources.

Aims

The overall goal of this study is to systematically investigate whether training on the mock MR scanner reduces the need for GA during MRI scans in children. There are three specific aims:

1. Determine whether pre-scan training allows children to have successful diagnostic MRI scans without general anesthesia.
2. Examine the effects of different types of pre-scan training on reducing anxiety and stress in children and their parents related to diagnostic MRI.
3. Determine whether mock scanner training can lower the age at which neuro-oncology patients are able to complete a full diagnostic MRI without anesthesia compared with historic controls.

Patient name, date of birth, and hospital identification number are necessary to perform chart review and access diagnostic images. All identifying information will be removed prior to data analysis.

The following data will be collected/recorded for each participant at enrollment:

1. Study number
2. Sex
3. Age at time of scan(s)
4. Type of diagnostic scans requested
5. Parent report on overall stress
6. Parent proxy measures of child stress/worry (PedsQL)
7. Parent predictions of child success on MRI
8. (Aim 3 only) Primary Oncology Diagnosis: i) Site ii) Histology
9. (Aim 3 only) Treatment mode i) Surgery ii) Chemotherapy iii) Radiotherapy

Training Sessions

For Aims 1 and 2, participants will be randomly assigned to one of three training groups. Group 1 will be sent links to online videos about MRI, audio files with scanner noises, and a children's book about MR scans, to prepare at home. Group 2 will receive training materials and visit the ACH to review them with the research team, but will not use the mock scanner. Group 3 will receive training materials and visit the ACH for training on the mock MR scanner. Visits to the mock scanner for Group 3 will include practice lying down, staying still, wearing headphones, and watching a movie on the mirror system. The Child Life Specialist will talk with the child and his/her family about the experience, and allow them up to 1 hour of practice time on the mock scanner.

For Aim 3, all participants will receive training on the mock scanner similar to group 3 with the difference being Child Life Specialists will utilize a goal based preparation of 3 X 20 minute sessions to coincide with other visits to the hospital.

All participants will be booked for one MR scan without GA and one with GA a week later in case the first scan fails.

The following data will be collected during/after training sessions:

1. Total time spent preparing (mock scanner or other)
2. Child's feelings of stress/worry before and after visit (PedsQL)
3. Head motion during mock MRI session (if applicable)

Diagnostic MRI Sessions

The following information will be recorded for each child's MRI scan:

1. Date of MRI.
2. Child's age at time of scanning.
3. Scan success without anesthesia (pass/fail)
4. Number of sequences requiring repeating
5. Total scan length (mins)
6. Sum of individual scan sequence times (mins)
7. Quality of images, as determined by a pediatric neuro-radiologist and graded as Excellent (no motion artifact ), Good (minimal motion artifact ); Acceptable (motion artifact; but satisfactory to answer the clinical question); Unacceptable (significant motion artifact ; unable to answer the clinical question)
8. Parent proxy measures of child stress ( PedsQL )
9. Child's stress/worry (PedsQL)
10. (Aims 1 and 2) Saliva sample to measure cortical and salivary alpha amylase before and after diagnostic MR scan

If images are deemed suitable for clinical diagnosis, the subsequent GA booking will be cancelled.

No raw images will be retained for any patients outside of their hospital record.

For Aim 3 prospective data, the above information will be recorded at each scanning session until the patient is able to complete the entire scan without anesthesia.

For Aim 3 retrospective data: The patient's hospital identification number will be used to identify MRI scans performed on that patient in the 3 years prior to the study. The MRI report will be cross referenced with the department of anesthesia electronic database to determine the date and thereby the age at which MRI without GA was able to be performed. In the case where the MRI report states that scan was performed under GA but no electronic record of GA is present the paper chart will be reviewed to determine if GA was performed. If The MRI scan report does not specify that GA was performed and an anesthesia record for the MRI exists then scan will be considered to have been performed under GA.

Statistical Plan

An ANOVA will be used to evaluate group differences on scanning success measures. Additional analyses will focus on correlations between scan successes and age, sex, measures of child/parent stress, cortisone, salivary alpha amylase, and training session compliance.

Aim 3 will also explicitly test differences in the mean age in months at which neuro-oncology patients were able to successfully complete the diagnostic MRI without anesthesia in the groups with and without mock scanner training. These will be compared utilizing T-test and Kaplan-Meier Analysis.

ELIGIBILITY:
Inclusion Criteria:

* Elective MRI scans
* No previous Diagnostic MRI without GA
* Would normally receive GA for diagnostic MRI
* No significant developmental delay
* Ability to understand English for groups 1,2 and 3.
* For neuro-oncology group: Ability of accompanying parent and/or child to communicate in English with regular exposure of the child to the English language
* For Neuro-oncology subgroup:a diagnosis of primary brain tumor under the care of neuro-oncology at Alberta Children's Hospital

Exclusion Criteria:

* Inability to understand consent form
* Urgent Scans (insufficient time to prepare)
* Previous diagnostic MRI without the need for general anesthesia
* Fast brain MRI (single sequence for sole purpose of determining size of cerebrospinal fluid (CSF) spaces)

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Success of Diagnostic Scan | Immediate: on the date of scheduled MRI
  Whether child is able to complete a diagnostic MRI scan without general anesthesia
Neuro-oncology Age of completion of MRI without GA | 3 years
  Determine the age at which neuro-oncology patients can complete a full diagnostic MRI without requiring general anesthesia

SECONDARY OUTCOMES:
Quality of scan Quality of MRI for diagnostic purposes | Immediate: on the date of scheduled MRI
  Ability to use scan for diagnostic purpose
Time taken to complete diagnostic MRI | Immediate: on the date of scheduled MRI
  Time in minutes
Number of scan sequences that require repeating | Immediate: on the date of scheduled MRI
  Number of scans sequences that need repeating
Childs feelings of stress | Immediate: on the date of scheduled MRI
  Using Peds QL child version and parent proxy version to quantify stress
Salivary stress hormone levels (cortisol & alpha amylase) | Immediate: on the date of scheduled MRI
  Salivary stress hormones will be measured for training groups 1,2 and 3
Compliance with training | 2 weeks
  recording the amount of time preparation took

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Lebel, PhD, Principal Investigator — catherine.lebel@albertahealthservices.ca
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnea-Goraly N, Weinzimer SA, Ruedy KJ, Mauras N, Beck RW, Marzelli MJ, Mazaika PK, Aye T, White NH, Tsalikian E, Fox L, Kollman C, Cheng P, Reiss AL; Diabetes Research in Children Network (DirecNet). High success rates of sedation-free brain MRI scanning in young children using simple subject preparation protocols with and without a commercial mock scanner--the Diabetes Research in Children Network (DirecNet) experience. Pediatr Radiol. 2014 Feb;44(2):181-6. doi: 10.1007/s00247-013-2798-7. Epub 2013 Oct 6. PMID 24096802
- [Background] de Bie HM, Boersma M, Wattjes MP, Adriaanse S, Vermeulen RJ, Oostrom KJ, Huisman J, Veltman DJ, Delemarre-Van de Waal HA. Preparing children with a mock scanner training protocol results in high quality structural and functional MRI scans. Eur J Pediatr. 2010 Sep;169(9):1079-85. doi: 10.1007/s00431-010-1181-z. Epub 2010 Mar 13. PMID 20225122
- [Background] Lueken U, Muehlhan M, Evens R, Wittchen HU, Kirschbaum C. Within and between session changes in subjective and neuroendocrine stress parameters during magnetic resonance imaging: A controlled scanner training study. Psychoneuroendocrinology. 2012 Aug;37(8):1299-308. doi: 10.1016/j.psyneuen.2012.01.003. Epub 2012 Feb 5. PMID 22309826
- [Background] Raschle NM, Lee M, Buechler R, Christodoulou JA, Chang M, Vakil M, Stering PL, Gaab N. Making MR imaging child's play - pediatric neuroimaging protocol, guidelines and procedure. J Vis Exp. 2009 Jul 30;(29):1309. doi: 10.3791/1309. PMID 19684560
- [Background] Sherman SA, Eisen S, Burwinkle TM, Varni JW. The PedsQL Present Functioning Visual Analogue Scales: preliminary reliability and validity. Health Qual Life Outcomes. 2006 Oct 4;4:75. doi: 10.1186/1477-7525-4-75. PMID 17020606
- [Background] Carter AJ, Greer ML, Gray SE, Ware RS. Mock MRI: reducing the need for anaesthesia in children. Pediatr Radiol. 2010 Aug;40(8):1368-74. doi: 10.1007/s00247-010-1554-5. Epub 2010 Feb 26. PMID 20186541
- [Background] Hallowell LM, Stewart SE, de Amorim E Silva CT, Ditchfield MR. Reviewing the process of preparing children for MRI. Pediatr Radiol. 2008 Mar;38(3):271-9. doi: 10.1007/s00247-007-0704-x. Epub 2007 Dec 15. PMID 18084752
- [Background] Pressdee D, May L, Eastman E, Grier D. The use of play therapy in the preparation of children undergoing MR imaging. Clin Radiol. 1997 Dec;52(12):945-7. doi: 10.1016/s0009-9260(97)80229-2. PMID 9413970
- [Background] de Amorim e Silva CJ, Mackenzie A, Hallowell LM, Stewart SE, Ditchfield MR. Practice MRI: reducing the need for sedation and general anaesthesia in children undergoing MRI. Australas Radiol. 2006 Aug;50(4):319-23. doi: 10.1111/j.1440-1673.2006.01590.x. PMID 16884416
- [Background] Tyc VL, Fairclough D, Fletcher B, Leigh L, Mulhern RK. Children's distress during magnetic resonance imaging procedures. Child Health Care. 1995 Winter;24(1):5-19. doi: 10.1207/s15326888chc2401_2. PMID 10142086